CLINICAL TRIAL: NCT05254041
Title: Pilot Study of Suction as a Mechanism of IUD Expulsion With Concomitant Menstrual Cup Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-4267
Record Dates: First submitted 2022-01-28; First posted 2022-02-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: IUD; Complications, Mechanical; Menstrual Cup

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mentrual Cup Removal (Other): Menstrual Cup Removal.
  Interventions: Other: Menstrual Cup Removal

INTERVENTIONS:
Other: Menstrual Cup Removal — Participants will be asked to remove Menstrual cup by breaking the seal.

SUMMARY:
This study will provide pilot data examining suction as a mechanism of IUD displacement with menstrual cup use. The investigator hypothesize that manufacturer-recommended menstrual cup insertion and removal by breaking the seal will result in 15% rate of IUD displacement/expulsion. The investigator will also use this data to explore variables associated with IUD displacement and menstrual cup use. By examining the role of suction as a possible mechanism of IUD displacement, this research will allow healthcare providers to better counsel patients who use IUDs regarding menstrual cup use. Having a better understanding of the mechanics of IUD displacement could lead to the development of strategies to prevent expulsion.

DETAILED DESCRIPTION:
Intrauterine devices (IUDs) are a commonly used, highly effective form of long-acting, reversible contraception in the United States (US). IUD expulsions, or displacement of the IUD from the top of the uterine cavity occur approximately 5% of the time but can have significant consequences for patients such as unintended pregnancy and further need for health care services and costs. Limited data suggests that menstrual cup use with an IUD in place may be associated increased risk of IUD expulsion. Menstrual cups such as the DivaCup are reusable collection devices that are an increasingly popular alternative to tampons or sanitary pads in the US; they are more cost effective and more environmentally sustainable. The cup is placed in the vagina to create a vacuum seal to prevent leakage. This seal or suction should be released before cup removal. Two plausible mechanisms have been suggested to explain IUD expulsion in the setting of menstrual cup use: the suction created by the cup displaces the IUD, or the IUD strings are inadvertently pulled on during cup removal. No studies have examined the mechanics of IUD displacement. Additionally, there are no formal recommendations guiding patients and providers about concomitant IUD and menstrual cup use, including expulsion risk or strategies to prevent expulsions. Data are needed to not only better understand the mechanisms of IUD displacement with menstrual cup use, but to better guide the many patients who use both.

This study will address this knowledge gap by performing an exploratory study of the IUD displacement with menstrual cup insertion and removal, specifically looking at suction as a mechanism. The investigator will enroll fifty women presenting for IUD removal. Women will be screened for eligibility and participants will be excluded if they are unable to place and remove a menstrual cup, do not have visible IUD strings on exam, have a silicone allergy or sensitivity, or have an experimental IUD. After a screening pelvic exam and transvaginal ultrasound to measure the distance of the IUD from the top of the uterine fundus, the participant will be asked to place a menstrual cup as suggested by the manufacturer. Participants will then be instructed to remove the menstrual cup by breaking the suction or seal. A repeat transvaginal ultrasound will be done to re-measure the IUD location and quantify any displacement. Participants who did not have complete IUD expulsion with the first cup placement and removal will be instructed to replace the cup and then remove the cup without breaking the seal.

This study will provide pilot data examining suction as a mechanism of IUD displacement with menstrual cup use. The investigator hypothesize that manufacturer-recommended menstrual cup insertion and removal by breaking the seal will result in 15% rate of IUD displacement/expulsion. The investigator will also use this data to explore variables associated with IUD displacement and menstrual cup use. By examining the role of suction as a possible mechanism of IUD displacement, this research will allow healthcare providers to better counsel patients who use IUDs regarding menstrual cup use. Having a better understanding of the mechanics of IUD displacement could lead to the development of strategies to prevent expulsion.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between the ages of 18-45
* Currently has an FDA approved IUD
* Present to CWHC for IUD removal

Exclusion Criteria:

* Known sensitivity or allergy to silicone
* known active vaginal infection (yeast, bacterial vaginosis, untreated sexually transmitted infection)
* IUD strings not visible
* Positive pregnancy test

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Limited to only females as IUDs are only approved for females
Enrollment: 80 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of IUD displacement with manufacturer-recommended menstrual cup insertion and removal | 12-18 months
  The rate of IUD displacement measured by the frequency of IUDs that shift >1cm after manufacturer-recommended menstrual cup insertion and removal.

SECONDARY OUTCOMES:
The rate of IUD displacement measured by the frequency of IUDs that shift >1cm after manufacturer-recommended menstrual cup insertion and removal followed by insertion and removal the menstrual cup without breaking the seal. | 12-18 months
  The rate of IUD displacement measured by the frequency of IUDs that shift >1cm after manufacturer-recommended menstrual cup insertion and removal followed by insertion and removal the menstrual cup without breaking the seal.

OTHER OUTCOMES:
III. The proportion of subjects who report pulling on the menstrual cup stem before breaking the seal. | 12-18 months
  The proportion of subjects who report pulling on the menstrual cup stem before breaking the seal.
III. The proportion of subjects who report feeling suction during menstrual cup removal. | 12-18 months
  The proportion of subjects who report feeling suction during menstrual cup removal.
III. The proportion of subjects who report palpating the IUD strings during menstrual cup removal. | 12-18 months
  The proportion of subjects who report palpating the IUD strings during menstrual cup removal.

CONTACTS AND LOCATIONS:
Overall Officials: Cara Clure, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Comprehensive Women's Health Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Daniels K, Daugherty J, Jones J, Mosher W. Current Contraceptive Use and Variation by Selected Characteristics Among Women Aged 15-44: United States, 2011-2013. Natl Health Stat Rep. 2015; 86:1-14. — https://pubmed.ncbi.nlm.nih.gov/26556545/
- See also: Daniels K, Abma JC. Current Contraceptive Status Among Women Aged 15-49: United States, 2017-2019. NCHS Data Brief. 2020:1-8. — https://pubmed.ncbi.nlm.nih.gov/33151146/
- See also: Kaiser Family Foundation. Intrauterine Devices (IUDs): Access for Women in the U.S. — https://www.kff.org/womens-health-policy/fact-sheet/intrauterine-devices-iuds-access-for-women-in-the-u-s/
- See also: U.S. Food and Drug Administration Prescribing Information: Mirena (levonorgestrel-releasing intrauterine system). Reference ID: 3837008. — https://www.accessdata.fda.gov/drugsatfda_docs/label/2020/021225s040lbl.pdf
- See also: U.S. Food and Drug Administration Prescribing Information: ParaGard (intrauterine copper contraceptive). Reference ID: 3321877. — https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/018680s069s070lbl.pdf
- See also: Teal SB, Turok DK, Chen BA, Kimble T, Olariu AI, Creinin MD. Five-Year Contraceptive Efficacy and Safety of a Levonorgestrel 52-mg Intrauterine System. Obstet Gynecol. 2019;133:63-70. — https://pubmed.ncbi.nlm.nih.gov/30531565/
- See also: Boortz HR, Margolis DJA, Ragavendra N, et al. Migration of intrauterine devices: radiologic findings and implications for patient care. Radiographics. 2012; 32:335-352. — https://pubmed.ncbi.nlm.nih.gov/22411936/
- See also: Madden T, McNicholas C, Zhao Q et al. Association with age and parity with intrauterine device explusion. Obstet Gynecol. 2014; 124: 718-726 — https://pubmed.ncbi.nlm.nih.gov/25198262/
- See also: Seale R, Powers L, Guiahi M, Coleman-Minahan K. Unintentional IUD expulsion with concomitant menstrual cup use: a case series. Contraception. 2019; 100: 85-87. — https://pubmed.ncbi.nlm.nih.gov/30981842/
- See also: Gilliam ML, Jensen JT, Eisenberg DL, Thomas MA, Olariu A, Creinin MD. Relationship of partity and prior cesarean delivery to levonorgestrel 52 mg intrauterine system expulsion over 6 years. Contraception. 2021; 22: 1-6. — https://pubmed.ncbi.nlm.nih.gov/33651995/
- See also: DivaCup®. 2021. Accessed date: 16 March 2021. — https://divacup.com/
- See also: Lunette®. /;2021. Accessed date: 16 March 2021. — https://store.lunette.com
- See also: Jones L. Why are menstrual cups becoming more popular? BBC news. Available at: https://www.bbc.com/news/business-45667020; 2018, Accessed date: 16 March 2021. — https://www.bbc.com/news/business-45667020
- See also: Schnyer AN, Jensen JT, Edelman A, Han L. Do menstrual cups increase risk of IUD expulsion? A survey of self-reported IUD and menstrual hygiene product use in the United States. Eur J Contracept Reprod Health Care. 2019; 24: 368-372 — https://pubmed.ncbi.nlm.nih.gov/31335218/
- See also: Long J, Schreiber C, Creinin MD, Kaneshiro B, Nanda K, Blithe D. Menstrual cup use and intrauterine device expulsion in a copper intrauterine device efficacy trial [OP01-1B]. Obstet Gynecol. 2020; 135:1S. — https://escholarship.org/uc/item/5kz1t720
- See also: Menstrual Cup Reviews. https://menstrualcupreviews.net/high-or-low-cervix/;2019. Accessed date: 16 March 2021 — https://menstrualcupreviews.net/high-or-low-cervix
- See also: Wiebe ER, Trouton KJ. Does using tampons or menstrual cups increase early IUD expulsion rates? Contraception. 2012; 86: 119-21. — https://pubmed.ncbi.nlm.nih.gov/22464406/
- See also: Lunette®. Can you use a menstrual cup with an IUD? https://store.lunette.com/blogs/news/can-you-use-menstrual-cup-with-iud; 2018. Accessed date: 16 March 2021. — https://store.lunette.com/blogs/news/can-you-use-menstrual-cup-with-iud
- See also: Kattan DR, Burkamn R. Overcoming LARC complications: 7 case challenges. OBG Management. 2017; 29:18-24. — https://www.mdedge.com/obgyn/article/126597/contraception/overcoming-larc-complications-7-case-challenges